CLINICAL TRIAL: NCT02012062
Title: Phase Ⅲ Study of Neoadjuvant TPF Chemotherapy Followed by Radiotherapy With Concurrent Nimotuzumab or Cisplatin for Locoregionally Advanced Nasopharyngeal Carcinoma (NPC).
Brief Title: Concurrent Nimotuzumab Versus Cisplatin With Radiotherapy for Locoregionally Advanced NPC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Fujian Province Tumor Hospital (Other); The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Lin Kong, Dr., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPC-IMRT-N
Record Dates: First submitted 2013-12-04; First posted 2013-12-16 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; Neoadjuvant chemotherapy; Concurrent chemotherapy; Nimotuzumab
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm Cisplatin (Active Comparator): Neoadjuvant TPF chemotherapy (docetaxel 75 mg/m2, cisplatin 75 mg/m2, 5-FU 2500 mg/m2 every 3 weeks for 3 cycles), followed by cisplatin 40 mg/m2/week in concurrent with IMRT
  Interventions: Drug: TPF neoadjuvant chemotherapy; Drug: Concurrent chemotherapy with cisplatin during radiotherapy; Radiation: Radical radiotherapy
- Arm Nimotuzumab (Experimental): Neoadjuvant TPF chemotherapy (docetaxel 75 mg/m2, cisplatin 75 mg/m2, 5-FU 2500 mg/m2 every 3 weeks for 3 cycles), followed by weekly nimotuzumab 200mg in concurrent with IMRT
  Interventions: Drug: TPF neoadjuvant chemotherapy; Drug: Concurrent nimotuzumab during radiotherapy; Radiation: Radical radiotherapy

INTERVENTIONS:
Drug: TPF neoadjuvant chemotherapy
Drug: Concurrent chemotherapy with cisplatin during radiotherapy
  Arms: Arm Cisplatin
Drug: Concurrent nimotuzumab during radiotherapy
  Arms: Arm Nimotuzumab
Radiation: Radical radiotherapy

SUMMARY:
The study is to evaluate whether concurrent nimotuzumab could decrease the severe acute treatment-related toxicities compared with concurrent chemoradiotherapy for locoregionally advanced NPC. Three hundreds and twenty patients will be recruited into this study.

DETAILED DESCRIPTION:
Scheme:

Eligible stage III and IVA/B NPC patients will first be stratified by institution, then randomized to 2 arms at 1:1 ratio.

- Arm Cisplatin:

Neoadjuvant TPF chemotherapy (docetaxel 75 mg/m2, cisplatin 75 mg/m2, 5-FU 2500 mg/m2 every 3 weeks for 3 cycles), followed by cisplatin 40 mg/m2/week in concurrent with IMRT

- Arm nimotuzumab:

Neoadjuvant TPF chemotherapy (docetaxel 75 mg/m2, cisplatin 75 mg/m2, 5-FU 2500 mg/m2 every 3 weeks for 3 cycles), followed by weekly nimotuzumab 200mg in concurrent with IMRT

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven poorly differentiated or undifferentiated carcinoma of the nasopharynx.
* Stage III and IVA/B NPC patients
* KPS >70
* Age between 18-70
* AGC > 2000, platelets > 100,000, AST or ALT<2 x upper normal, serum creatinine<1.5mg/dl, creatinine clearance >50ml/min

Exclusion Criteria:

* Histology other than poorly differentiated or undifferentiated carcinoma, including keratinized squamous cell carcinoma.
* Evidence of metastases (below the clavicle or distant) by clinical or radiographic examinations.
* Initial surgical treatment excluding diagnostic biopsy of the primary site or neck disease.
* Patients with simultaneous or prior malignancy (not include basal cell carcinoma of skin)
* Prior radiation treatment to the head and neck or any prior chemotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (severe radiation-induced skin and mucosal toxicities) | From Day 1 to Day 90 of radiotherapy

SECONDARY OUTCOMES:
PFS | 3 years
OS | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China